CLINICAL TRIAL: NCT02690935
Title: Randomized, Double-blind, Placebo-controlled Study to Measure 2L®ALERG (Homeopathic Drug) Efficacy on Symptoms of Allergic Rhinitis and Allergic Rhinoconjunctivitis in Patients With a Seasonal Allergy to Grass Pollen
Brief Title: Efficacy of 2LALERG (Homeopathic Drug) in Allergic Rhinitis Related to Grass Pollen
Acronym: LLB-2016-01
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Labo'Life (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LLB-2016-01
Record Dates: First submitted 2016-02-17; First posted 2016-02-24 (Estimated); Results first posted 2017-12-15 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2017-10

CONDITIONS: Seasonal Allergy
Keywords: grass pollen; homeopathy; placebo; quality of life
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — Immunotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2LALERG (Experimental): Interleukin 1: 17 CH Interleukin 4: 17-27 CH Interleukin 5: 17 CH Interleukin 6: 17 CH Interleukin 10: 17 CH Interleukin 12: 9 CH Interleukin 13: 17 CH Tumor Necrosis Factor Alpha: 17 CH Transforming Growth Factor Beta: 5 CH Pulmo histaminum: 15 CH SNA-HLA-II: 18 CH
  Impregnated on lactose saccharose globules (380 mg/capsule)
  Interventions: Drug: 2LALERG
- Placebo (Placebo Comparator): Non-impregnated lactose saccharose globules (380 mg/capsule)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 2LALERG — Homeopathic drug
  Other Names: Immunotherapy
  Arms: 2LALERG
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The primary objective of this study is to demonstrate the superiority of 2L®ALERG over placebo in terms of efficacy on the symptoms of allergic rhinitis and allergic rhinoconjunctivitis in patients with seasonal allergy to grass pollen, corrected according to rescue medication intake. The secondary objectives are to compare the allergy symptoms, the rescue medication intake, the quality of life and the safety in patients treated with 2L®ALERG or with a placebo.

This is a multicentre, randomized, double-blind, two-parallel group, interventional placebo-controlled study with a notified homeopathic medication, marketed since 2002.

Fifty patients will be recruited per group to achieve 40 cases completed per group, i.e., a total of 100 patients included for 80 cases completed.

Screening will be done before the peak of pollination and the treatment will be set up two months before traditional pollen peak, then visits at 3 months and 6 months, or end of the peak.

The treatment will consist of 1 capsule daily, fasting morning, following the numerical order of 1 to 10 capsules for 6 months.

The placebo will have the same form, colour, taste and aspect. The allowed concomitant treatments are the already established treatments for associated pathologies not liable to have an impact on the proper conduct of the study and the rescue medications allowed in the first-line adjuvant treatment (oral or topical antihistamines [nasal or eye] and eye cromoglycate, topical nasal corticosteroids [in case of failure or insufficiency of those above]).

The prohibited treatments are the oral or injectable corticosteroids and the anti-leukotrienes.

DETAILED DESCRIPTION:
The primary objective of this study is to demonstrate the superiority of 2L®ALERG over placebo in terms of efficacy on the symptoms of allergic rhinitis and allergic rhinoconjunctivitis in patients with seasonal allergy to grass pollen, corrected according to rescue medication intake. The secondary objectives are to compare the allergy symptoms, the rescue medication intake, the quality of life and the safety in patients treated with 2L®ALERG or with a placebo.

This is a multicentre, randomized, double-blind, two-parallel group, interventional placebo-controlled study with a notified homeopathic medication, marketed since 2002.

Fifty patients will be recruited per group to achieve 40 cases completed per group, i.e., a total of 100 patients included for 80 cases completed.

Screening will be done before the peak of pollination and the treatment will be set up two months before traditional pollen peak, then visits at 3 months and 6 months, or end of the peak.

The treatment will consist of 1 capsule daily, fasting morning, following the numerical order of 1 to 10 capsules for 6 months.

The placebo will have the same form, colour, taste and aspect. The allowed concomitant treatments are the already established treatments for associated pathologies not liable to have an impact on the proper conduct of the study and the rescue medications allowed in the first-line adjuvant treatment (oral or topical antihistamines [nasal or eye] and eye cromoglycate, topical nasal corticosteroids [in case of failure or insufficiency of those above]).

The prohibited treatments are the oral or injectable corticosteroids and the anti-leukotrienes.

The following demographic data will be collected during the first visit: date of birth, gender, ethnic group, weight, height, smoking habits and alcohol use status.

Medical history, treatment history, concomitant treatments and patient's physical examination will also be documented during V0.

The allergy must be confirmed by positive skin test and/or the presence of IgE for grasses (prick test defined as positive if higher than or equal to half the negative control; IgE are positive if at least class 3 (≥ 3.5 kU / L); these tests must have been made at the latest during the first visit.

A patient diary will be given to each patient:

* For evaluation of the total 5 symptoms score T5SS and rescue medication RS, it is essential that patients note every day the symptoms (sneezing, rhinorrhoea, nasal pruritus, itching and/or eye tearing and nasal obstruction) intensity, and the rescue medications, in their patient diary.
* It is also essential that the patient takes note every day of his/her QoL by filling in three questions included in his/her diary card: Did you sleep well? - Can you work normally? - How do you feel?
* It is also imperative that patients note the date of the start of treatment and the date of onset of symptoms.

This patient diary will be given to the patient at each visit, and will be brought back at the next visit, it will be reviewed and validated by the investigator and will be part of the Case Report Form.

All relevant (related to allergy) concomitant medications taken by the patient during the study period will be recorded at each visit in the CRF.

The AEs and SAEs will be recorded at V1 and V2 in order to assess safety.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years, male and female
* Woman of childbearing age using effective contraceptive means
* Patient having the faculties to understand and respect the constraints of the study
* Symptomatic since at least two seasons and confirmed by positive skin test and/or the presence of IgE for grasses (prick test defined as positive if higher than or equal to half the negative control; IgE positive if at least class 3 (≥ 3.5 kU / L); these tests must have been performed at the latest at the first screening visit
* Signature of the Informed Consent Form

Exclusion Criteria:

* Pregnant woman or woman wishing to become pregnant
* Breastfeeding woman
* Patient with an acute exacerbation of allergic rhinitis
* Patient with uncontrolled asthma
* Immunotherapy received within the last two years
* Patient with a known lactose intolerance
* Patient who participated in a clinical study in the previous three months
* Patient who is not sufficiently motivated to engage on a follow-up period of 6 months or more, unable to complete the patient diary, or likely to travel or to move before the end of the study,
* Patient taking nasal or bronchial inhaled corticosteroids on a long term basis (intermittent consumption during the season is permitted provided it is mentioned in the patient's records)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2016-03; Primary Completion 2017-04-07 (Actual); Study Completion 2017-04-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane Heijmans, MD, Principal Investigator — ResearchLink
Locations (1):
- ResearchLink, Linkebeek, Belgium

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first patient was enrolled in the study on 05 March 2016 and the last study visit was on 29 November 2016.
Groups:
- 2LALERG: Interleukin 1: 17 CH Interleukin 4: 17-27 CH Interleukin 5: 17 CH Interleukin 6: 17 CH Interleukin 10: 17 CH Interleukin 12: 9 CH Interleukin 13: 17 CH Tumor Necrosis Factor Alpha: 17 CH Transforming Growth Factor Beta: 5 CH Pulmo histaminum: 15 CH SNA-HLA-II: 18 CH
  Impregnated on lactose saccharose globules (380 mg/capsule)
  2LALERG: Homeopathic drug
Period: Overall Study
Arm/Group | 2LALERG | Placebo
Started | 51 (Count of participants) | 51 (Count of participants)
Completed | 51 (Count of participants) | 51 (Count of participants)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: No difference
Groups:
- Total: Total of all reporting groups
Arm/Group | 2LALERG | Placebo | Total
Number analyzed (Participants) | 51 | 51 | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.5 (14.5) | 40.7 (15.1) | 40.1 (14.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 26 | 49
  Male | 28 | 25 | 53
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 51 | 51 | 102
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Belgium | 51 | 51 | 102

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve [AUC](Total Score of Symptoms Taking Into Account the Total 5 Symptom Score (T5SS) and Consumption of Rescue Medications (RM) on the Y-axis, and Time on X Axis)
Description: Area under the curve [AUC] (total score of symptoms taking into account the Total 5 Symptom Score (T5SS) and consumption of rescue medications (RM) on the Y-axis versus time on X axis). T5SS was the sum of the 5 individual scores (min-max=0-15). It was corrected each day as a function of consumption of rescue medications (RM): oral antihistamine (+2 points), local treatment (nasal or eye; +1 point), ocular cromoglycate (+1 point) and nasal topical corticosteroids (+1 point). An increase in the total corrected score was considered as a worsening of the allergic symptoms.
Time Frame: Up to Month 6 (end of pollen season)
Population: ITT population
Measure: Mean (Standard Deviation); unit: T5SS score corrected with RM * day
Arm/Group | 2LALERG | Placebo
Number analyzed (Participants) | 49 | 47
T5SS score corrected with RM * day | 2.76 (1.89) | 2.97 (2.48)
Statistical Analysis 1: Comparison: 2LALERG vs Placebo; H0: The efficacy of 2LALERG and placebo are similar H1: The efficacy of 2LALERG and placebo are different; Test type: Superiority; p = 0.642, t-test, 2 sided — No adjustment of the p-value

2. Secondary Outcome: Quality of Life During the Whole Period of Observation
Description: This is the mean of the score to 3 daily quality of life questions: 1) Did you sleep well (0 to 3), 2) Are you able to work (0 to 3), 3) How do you feel today (0 to 3). The minimum daily score is 0 (good quality of life) and the maximum is 9 (bad quality of life). The mean of the daily scores was calculated over the whole period of observation (up to 6 months) for each patient.
Time Frame: QoL scores were assessed daily for up to 6 months
Population: ITT population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 2LALERG | Placebo
Number analyzed (Participants) | 49 | 47
units on a scale | 0.84 (0.88) | 0.81 (0.81)
Statistical Analysis 1: Comparison: 2LALERG vs Placebo; H0: 2LALERG and placebo have the same effect on the quality of life H1: 2LALERG and placebo do not have the same effect on the quality of life; Test type: Superiority; p = 0.829, t-test, 2 sided — No adjustment for multiplicity

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | 2LALERG | Placebo
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/51
Serious Adverse Events (participants affected / at risk) | 1/51 | 2/51
Other Adverse Events (participants affected / at risk) | 7/51 | 7/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2LALERG (N=51) | Placebo (N=51)
Cocaine abuse (Psychiatric disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Transient ischemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2LALERG (N=51) | Placebo (N=51)
Enteritis (Gastrointestinal disorders) | 3 (3) | 1 (1)
Bronchitis (Infections and infestations) | 3 (3) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)

LIMITATIONS AND CAVEATS:
1. Allergy cases were mainly prevalent and chronic.
2. Many concomitant drugs were taken
3. Patients were older in this trial compared to Van der Brempt et al. (2011)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2016-02-04): https://cdn.clinicaltrials.gov/large-docs/35/NCT02690935/Prot_002.pdf
  • Statistical Analysis Plan (2016-02-29): https://cdn.clinicaltrials.gov/large-docs/35/NCT02690935/SAP_003.pdf